CLINICAL TRIAL: NCT00817908
Title: Quantiferon - CMV and the Prediction of CMV Infection In High Risk Solid Organ Transplant Recipients
Brief Title: Quantiferon - Cytomegalovirus (CMV) and the Prediction of CMV Infection In High Risk Solid Organ Transplant Recipients
Status: Completed | Type: Observational
Sponsor: University of Alberta (Other)
Responsible Party: Principal Investigator, Deepali Kumar, Assistant Professor of Medicine, University of Alberta
Other Study IDs: 7267
Record Dates: First submitted 2008-10-15; First posted 2009-01-07 (Estimated); Last update posted 2012-04-23 (Estimated); Status verified 2012-04

CONDITIONS: Cytomegalovirus Infection
Keywords: liver transplant; lung transplant; kidney transplant; heart transplant; CMV CMI; Transplant
MeSH Terms: conditions — Cytomegalovirus Infections

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- 1: Patients at high risk for CMV infection (CMV serostatus: D+/R-) who are expected to receive three months of antiviral prophylaxis.

SUMMARY:
Cytomegalovirus (CMV) is a common cause of illness in patients who have undergone a transplant. Serious infections due to CMV can affect many parts of the body including the lungs, the gut, and the liver. Since transplant recipients are at risk for CMV or have evidence of infection with CMV, they are given an antiviral drug (usually ganciclovir or valganciclovir). Despite this, there are a chance that CMV infection may cause problems in the future. The purpose of this study is to assess how well patients'immune systems responds to the CMV virus, so that in the future it may be possible to predict which patients are at highest risk of CMV.

DETAILED DESCRIPTION:
CMV is the most common viral infection after solid organ transplantation (SOT) and is associated with significant morbidity1. Without prophylaxis, most CMV disease occurs in the first 3 months post-transplant during the period of intense of immunosuppresion.2 SOT recipients at the greatest risk are those that are seronegative recipients of organs from seropositive donors (CMV D+/R-).3, 4 Antiviral agents have proven to be useful in the prevention of CMV infection and disease in SOT recipients, including the high-risk D+/R- patients.5-9 Upon completion of prophylaxis however, CMV infection and disease occurs in about 50% and 25-30% respectively of D+/R- SOT recipients within the first year after transplant [30% rate of investigator treated CMV disease in PV16000].9 The incidence of CMV infection following prophylaxis in D+/R- lung transplant recipients may be as high as 80%.10 As CMV disease occurring after prophylaxis will continue to impact morbidity and mortality in SOT recipients, it would be desirable to be able to predict which patient will develop this complication. Currently, there are no reliable methods that are routinely available to predict the risk of CMV infection or disease in an individual patient. CMV viral load testing after prophylaxis in D+/R- patients has been shown to have poor predictive value for subsequent CMV disease.11 CMV serology (a measure of humoral immunity) was also shown to be only of marginal use in predicting the risk of late onset disease.12 Cell mediated immunity (CMI) is known to be more important than humoral immunity in controlling CMV infection. CMV infection elicits a strong virus specific CD4+ and CD8+ T-cell response. CD8+ T-cell responses to the virus often contain multiple antigen-specific reactivities including to viral pp65 or IE-1 antigens as well as pp50, glycoprotein B, and IE-2 and other antigens.13 CD4+ T cells also play a part in CMV control via promotion of priming, expansion and maintenance of CD8+ CMV-specific CTLs.14 Measuring an individual's CMI response to CMV may be a useful predictor of the risk of CMV infection or disease after prophylaxis. Patients with a poor CMI response (especially a poor CD8+ T-cell response) could then be targeted with longer courses of antiviral prophylaxis.

Cell mediated immunity testing Most of the previous studies have focused on CTL responses to the CMV phosphoprotein pp65.15-17 However, since CD8+ T-cell responses to CMV often contain multiple antigen-specific reactivities, measurement of CMI using epitopes restricted to a single protein may not yield adequate results. In conjunction with Dr. Rajiv Khanna (Queensland Institute of Medical Research, Australia), and Cellestis Ltd (Sydney, Australia), we have done preliminary validation and assessment of a CMI (Quantiferon-CMV) assay in which we measure the IFN-γ responses to a range of T-cell epitopes of CMV viral proteins including pp65, pp50, the glycoprotein gB, and the immediate early IE-1 antigen that are specific for a wide range of HLA class I specificities [See Appendix Table 1]. The assay employs a peptide pool for stimulation of whole blood and is suitable for routine clinical use and evaluation in multicenter studies.

The Quantiferon-CMV assay has been compared to an ELISPOT assay in a study involving 37 healthy volunteers and 25 SOT recipients.18 In this study, the Quantiferon-CMV assay was at least as sensitive as the ELISPOT for some CMV epitopes, and more sensitive for other CMV epitopes. In addition, the Quantiferon-CMV results highly correlated with the CMV serostatus, in both healthy volunteers and transplant recipients. In another study,19 the Quantiferon-CMV assay was used in HIV-infected individuals with and without a history of CMV disease. The CMV specific immune response measured by the Quantiferon-CMV assay was higher in patients without a history of CMV disease, suggesting that a positive result of the Quantiferon-CMV may predict the likelihood for developing a protective immune response against CMV.

ELIGIBILITY:
Inclusion Criteria:

Male or female patients who fulfill the following criteria are eligible for inclusion.

* CMV D+/R- liver, kidney, heart, pancreas, lungor combined transplant recipients
* All eligible patients must be scheduled to receive 3 months of either valganciclovir, oral ganciclovir, or intravenous ganciclovir prophylaxis.
* Able to give written informed consent
* Are willing and able to comply with the protocol
* Age >=18 years

Exclusion Criteria:

- Patient unwilling or unable to give informed consent

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: The study will aim to enrol 120 D+/R- transplant patients.
Sampling Method: Probability Sample
Enrollment: 131 (Actual)
Dates: Start 2008-05; Primary Completion 2012-03 (Actual); Study Completion 2012-04 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Atul Humar, MD, Principal Investigator — University of Alberta
Locations (1):
- University of Alberta Hospital, Edmonton, Alberta, Canada

REFERENCES:
- [Background] Razonable RR, Rivero A, Rodriguez A, Wilson J, Daniels J, Jenkins G, Larson T, Hellinger WC, Spivey JR, Paya CV. Allograft rejection predicts the occurrence of late-onset cytomegalovirus (CMV) disease among CMV-mismatched solid organ transplant patients receiving prophylaxis with oral ganciclovir. J Infect Dis. 2001 Dec 1;184(11):1461-4. doi: 10.1086/324516. Epub 2001 Oct 23. PMID 11709790
- [Background] Lowance D, Neumayer HH, Legendre CM, Squifflet JP, Kovarik J, Brennan PJ, Norman D, Mendez R, Keating MR, Coggon GL, Crisp A, Lee IC. Valacyclovir for the prevention of cytomegalovirus disease after renal transplantation. International Valacyclovir Cytomegalovirus Prophylaxis Transplantation Study Group. N Engl J Med. 1999 May 13;340(19):1462-70. doi: 10.1056/NEJM199905133401903. PMID 10320384
- [Background] Flechner SM, Avery RK, Fisher R, Mastroianni BA, Papajcik DA, O'Malley KJ, Goormastic M, Goldfarb DA, Modlin CS, Novick AC. A randomized prospective controlled trial of oral acyclovir versus oral ganciclovir for cytomegalovirus prophylaxis in high-risk kidney transplant recipients. Transplantation. 1998 Dec 27;66(12):1682-8. doi: 10.1097/00007890-199812270-00019. PMID 9884259
- [Background] Paya C, Humar A, Dominguez E, Washburn K, Blumberg E, Alexander B, Freeman R, Heaton N, Pescovitz MD; Valganciclovir Solid Organ Transplant Study Group. Efficacy and safety of valganciclovir vs. oral ganciclovir for prevention of cytomegalovirus disease in solid organ transplant recipients. Am J Transplant. 2004 Apr;4(4):611-20. doi: 10.1111/j.1600-6143.2004.00382.x. PMID 15023154
- [Derived] Manuel O, Husain S, Kumar D, Zayas C, Mawhorter S, Levi ME, Kalpoe J, Lisboa L, Ely L, Kaul DR, Schwartz BS, Morris MI, Ison MG, Yen-Lieberman B, Sebastian A, Assi M, Humar A. Assessment of cytomegalovirus-specific cell-mediated immunity for the prediction of cytomegalovirus disease in high-risk solid-organ transplant recipients: a multicenter cohort study. Clin Infect Dis. 2013 Mar;56(6):817-24. doi: 10.1093/cid/cis993. Epub 2012 Nov 29. PMID 23196955